CLINICAL TRIAL: NCT06626269
Title: Identification of Innovative Biomarkers Related to the Immune System or Tumor Microenvironment to Promote the Efficacy of Immunotherapies
Acronym: HORIZON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023/841
Record Dates: First submitted 2024-10-02; First posted 2024-10-03 (Actual); Last update posted 2025-06-20 (Actual); Status verified 2025-06

CONDITIONS: Advanced Digestive Cancer; Advanced Gynecologic Cancer
Keywords: biomarker; immunology; gynecologic cancer; digestive cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- blood test (Experimental): In cohort A: patients with advanced digestive or gynecological cancers eligible to immunotherapies.
  In cohort B: patients with advanced digestive or gynecological cancers eligible to treatment without immunotherapy.
  In cohort C: patients with advanced digestive or gynecological cancers eligible to surgery of metastasis after chemotherapy.
  Interventions: Diagnostic Test: Blood sample; Other: Tumor tissue

INTERVENTIONS:
Diagnostic Test: Blood sample — In cohort A: 3 or 4 blood samples (for plasma and PBMC collection) : at baseline (before immunotherapy initiation); at 3 months ; at 12 months; on case of severe or unexpected toxicity.
  In cohort B: 3 blood sampes (for plasma and PBMC collection): at baseline (before treatment initiation); at 3 months ; at 12 months
  In cohort C: 2 blood samples (for plasma and PBMC collection) : at baseline (at the time of surgery); at 3 months (after surgery)
Other: Tumor tissue — Cohort A and B: 1 tumor block in paraffin at diagnosis + 1 tumor block in paraffin at progression (optional) Cohort C: Fresh tumoral tissue fragments for TIL and CAF + 1 tumor block in paraffin at time of surgery.

SUMMARY:
The immune system may be involved in the recognition and destruction of tumor cells or cells undergoing transformation. It is also currently accepted that the quality of immune responses can influence the evolution of cancers after chemotherapy.

In this context, it is possible to assess the presence of specific T cells in patients' blood and to correlate the presence of specific memory lymphocytes with the quality of long-term clinical protection.

The analysis of immune responses can also be based on i) analysis of the tumor microenvironment (analysis of surgical samples or biopsies) or ii) analysis of molecules secreted in plasma.

Today, the immunotherapies can generate clinical responses in several cancers (for 15 to 25% of patients with melanomas, bladder, lung, kidney or gastric cancers). But the development of these drugs raises two unresolved questions: i) what immunological parameters predict the efficacy of these treatments? ii) why do some cancers remain refractory to the efficacy of these immunomodulatory drugs? It is therefore necessary to identify biomarkers for prognostic stratification and monitoring of patients treated by immunotherapy.

The primary objective of our research team is to identify biomarkers related to the immune system or tumor microenvironment in order to better define patient eligibility criteria for immunotherapy strategies.

ELIGIBILITY:
INCLUSION CRITERIA:

General inclusion criteria:

* Patients ≥ 18 years old
* more than 6 months of life expectancy as assessed by the investigator
* Performance status ECOG 0 ; 1 or 2
* Patient affiliated to or beneficiary of French social security system
* Informed consent of the subject to participate in the study

Specific eligibility criteria:

- Cohort A [Patients with advanced digestive or gynecological cancers eligible to immunotherapies]: Patients with locally advanced or metastatic digestive or gynecological cancers A1: hepatocellular carcinoma eligible to immunotherapy ± antiangiogenic A2: biliary tract carcinoma eligible to chemo-immunotherapy A3: oesogastric carcinoma eligible to chemo-immunotherapy A4: other digestive localizations eligible to immunotherapy (anti-PD1/PDL1 ± anti-CTLA4) ± chemotherapy A5: gynecological cancers eligible to chemo-immunotherapy

- Cohort B [Patients with advanced digestive or gynecological cancers eligible to chemotherapy or targeted therapy without immunotherapy]: Patients with locally advanced or metastatic digestive or gynecological cancers B1: hepatocellular carcinoma eligible to antiangiogenic or chemotherapy B2: biliary tract carcinoma eligible to chemotherapy B3: oesogastric carcinoma eligible to chemotherapy B4: other digestive localizations eligible to chemotherapy and/or targeted therapy B5: gynecological cancers eligible to chemotherapy and/or targeted therapy

- Cohort C [Patients with advanced digestive or gynecological cancers eligible to surgery of metastasis after chemotherapy]: Patients with liver metastasis of colorectal cancer or peritoneal metastasis of ovarian cancer eligible to surgical resection

EXCLUSION CRITERIA :

General exclusion criteria:

* Patient under guardianship, curatorship or under the protection of justice
* Patient with any medical or psychiatric condition or disease, which would make the patient inappropriate for entry into this study
* Patient unlikely to cooperate with the study and/or poor cooperation anticipated by the investigator
* Patient without health insurance
* Pregnant women
* Subject within the exclusion period of another study or planned by the national volunteer file

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
for cohorts A and B: Progression free survival (PFS) at 6 months post treatment initiation | 6 months post treatment initiation
  Progression free survival (PFS) at 6 months post treatment initiation, defined as:
  * non progressive alive patients: if patients are alive without progression in the 6 months from the date of treatment initiation
  * or progressive or death patients: if patients are identified with a progression or a death in the 6 months from the date of treatment initiation
  * patients without progression or death and with follow up bellow than 6 months are not assessable for PFS status at 6 months Progression-free survival (PFS): defined as the delay from the date of treatment initiation to the disease progression or death from any cause whichever occurs first. Alive patient without progression will be censored at last radiological evaluation available showing no progression.
For cohort C: Relapse free survival (RFS) at 6 months after surgery of metastases | 6 months after surgery of metastases
  RFS: defined as the delay from the date of surgery of metastases to the disease relapse or death from any cause whichever occurs first. Alive patient without relapse will be censored at last radiological evaluation available showing no relapse.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - University Hospital of Besançon, Besançon
  - Georges François Leclerc center, Dijon

IPD SHARING:
Plan to Share IPD: No